CLINICAL TRIAL: NCT02923999
Title: Phase I Dose Escalation Trial to Evaluate Safety and Reactogenicity of Single IV Administration of P2G12
Brief Title: Study of Single IV Administration of P2G12
Acronym: FuturePharma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14.0231; 2016-001817-25 (EudraCT Number)
Record Dates: First submitted 2016-08-10; First posted 2016-10-05 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: HIV Infection
Keywords: HIV; MAB; PLANT
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose cohort 1 (Experimental): P2G12 0.125g
  Interventions: Drug: P2G12 Dose Cohort 1
- Dose cohort 2 (Experimental): P2G12 0.25g
  Interventions: Drug: P2G12 Dose Cohort 2
- Dose cohort 3 (Experimental): P2G12 0.5g
  Interventions: Drug: P2G12 Dose Cohort 3

INTERVENTIONS:
Drug: P2G12 Dose Cohort 1 — single dose of intravenous infusion: 0.125g of the P2G12 human monoclonal antibody
  Other Names: human monoclonal antibody
  Arms: Dose cohort 1
Drug: P2G12 Dose Cohort 2 — single dose of intravenous infusion: 0.25g of the P2G12 human monoclonal antibody
  Other Names: human monoclonal antibody
  Arms: Dose cohort 2
Drug: P2G12 Dose Cohort 3 — single dose of intravenous infusion: 0.5g of the P2G12 human monoclonal antibody
  Other Names: human monoclonal antibody
  Arms: Dose cohort 3

SUMMARY:
A randomised phase I trial of a monoclonal antibody which neutralises HIV-1 (P2G12) to be given as a single intravenous infusion to healthy human volunteers to assess the safety and reactogenicity

DETAILED DESCRIPTION:
Study disease:

In 2014 it was estimated that 36.9 million people worldwide were living with HIV and since the beginning of the epidemic, about 36 million have died of HIV.

There are many research strategies underway to try to reduce the devastating effects of this disease and to prevent onward transmission, and it is likely that a range of these used simultaneously will be required to bring the epidemic under control. These include the development of a vaccine, microbicide, antiviral treatment and agents used in prevention. Amongst these, a HIV neutralising antibody that is safe when infused intravenously could play an important role either in post exposure, or when HIV is driving an aggressive disease and there is a need to lower the viral load abruptly or when mothers present in labour with high viral loads.

The clinical advancement of monoclonal antibodies has been hampered by the inability to manufacture the specific recombinant proteins with a system that would be scalable for the global market. There is also a valid perception that even if manufacturing was possible, it would be at a totally unaffordable cost. Thus, neutralising monoclonal antibodies such as MAbs b12 have only reached efficacy studies in rhesus macaques. In the case of monoclonal antibodies it is generally believed that a cocktail of at least 3 antibodies would be necessary to avoid viral escape, thereby potentially tripling the cost of a product, as compared with a conventional single monoclonal antibody therapeutic. It is clear that in order to progress these promising anti-HIV monoclonal antibodies, new methods of manufacture need to be developed.

Investigational Medicinal Product (IMP):

P2G12 is a human IgG1 class monoclonal antibody (MAb) which has been expressed in tobacco plants (referred to as "P2G12" to indicate plant origin). The parent molecule ("2G12") is one of a handful of MAbs with potent neutralising activity against HIV and has been produced by CHO cell fermentation (referred to as "C2G12" to indicate CHO-cell origin). A number of studies have demonstrated that passively infused monoclonal antibodies can protect against an intravenous challenge by the infectious SHIV reagent in rhesus macaques. Furthermore, HIV neutralising MAbs can affect transmission and subsequent disease course after vaginal SHIV-challenge in macaques In studies in humans, the MAb C2G12 was safe after repeated intravenous infusions to asymptomatic HIV-1-infected individuals . Similarly, another MAb 4E10 was safe after intravenous infusions, alone and in combination with other MAbs including C2G12, to HIV-1-infected individuals These studies prepared the way for the introduction of these MAbs for human immunoprophylaxis against HIV infection and indeed new generation anti-HIV MAbs are currently being advanced in prophylactic and therapeutic children and adult clinical trials with children and adults With respect to the MAb 2G12, in a number of human clinical trials, 4 to 16 infusions of C2G12 were given in doses ranging from 0.5g to 1g alone or in combination with other MAbs. The safety results from these studies were reassuring with minimal adverse drug reactions observed. Those that were reported were of myalgia and arthralgia. In a recently conducted study, P2G12 was safe to use when administered intravaginally at a concentration of 7, 14 and 28mg/ml.

Pre-clinical toxicity studies of IV use (bolus) of P2G12 were completed on rats at doses of 7 and 35mg/kg (equivalent to 490mg and 2.45g for a 70Kg human respectively). No adverse events were observed up to 14 days post-administration, no safety concerns were raised.

Study design:

This will be a phase 1, randomised, single blinded dose escalation study in healthy adult volunteers. There will be three groups of 6 volunteers receiving increasing doses of the MAb. 0.125g dose group , the 0.25g dose group and the 0.5g dose group The volunteers will be followed up for 3 months post dose when safety and immunogenicity will be assessed.

Prior to any study specific procedures, each suitable participant will be given written information about the planned procedures and schedule. Each volunteer will be provided sufficient time to consider participation in the study. Any questions about the study will be answered by trained personnel. If the volunteers are still willing and interested they will be asked to sign the informed consent form (ICF). Participants will be advised that they are under no obligation to enter the trial and that they can withdraw at any time during the trial, without having to give a reason.

A copy of the signed ICF along with a copy of the most recent approved Patient Information Sheet (PIS) will be given to the study participant. An original signed & dated consent form will be retained in the medical notes (if available) or trial notes where medical notes are unavailable and a copy will be placed in the ISF.

To ensure informed consent, volunteers will go through the following processes in detail with a member of the study team:

1. Pre-HIV risk assessment and discussion
2. Safe sex counselling
3. That it is unknown whether or not the study vaccine will protect against HIV infection
4. The level of care that will be made available to them should they be found to be HIV infected at any time during their participation in the study, including the screening period
5. That they, or their partner should continue to use a reliable form of contraception for 14 days prior to the immunisation period and for 4 months afterwards
6. That they should continue to use condoms with sexual partners whose HIV status is not known
7. Risk assessment and discussion of intravenous infusions

After ICF has been collected, assessments and investigations will be undertaken according to the visit schedule.

Participants will be required to make a minimum of 8 scheduled outpatient visits over the course of 20 weeks.

Following informed consent at the screening visit, demographics, medical history, information about contraceptive practices and concomitant medication will be collected and safe sex consultation will take place. Height, weight and temperature will be recorded and full physical examination will be performed, vital signs and ECG will be recorded.

Peripheral blood will be collected and the following will be assessed:

* Hb, total WBC, neutrophils, lymphocytes and platelets
* Clotting screen
* creatinine, total bilirubin, alkaline phosphatase, AST, ALT and glucose
* serology for HBV (hepatitis B surface antigen), HCV (hepatitis C antibody) and HIV-1/HIV-2 (4th generation HIV antibody/antigen test) Urinalysis using a dipstick for protein, ketones, blood, leukocyte esterase, and nitrites and urine test to exclude pregnancy will be tested.

Results of the assessments taken place prior to administration of the IMP will be considered as baseline values.

Peripheral blood for serum will be collected for immunogenicity testing.

Medical report will be requested from the volunteer's GP to confirm eligibility.

As soon as the medical report is received and all required test results are available, this will be reviewed and eligibility signed off by the PI.

The participant will then be invited to receive the IMP on a mutually agreeable date

A simple randomisation schedule for each dose cohort will be generated using the web service. Infusion will be administered intravenously using an infusion pump. Participants will be blind to dose of IMP.

All patients will be given a study specific 24hrs emergency contact card with out of hours contact details in case of emergency.

Dosing visit:

P2G12 4mg/ml in sodium Chloride 0.9% w/v represented as sodium chloride 0.9% w/v to be administered over a total infusion period of 30 minutes. P2G12 infusions are clear solutions, this will allow single blinding.

The infusions will be delivered over 30 minutes with continuous monitoring throughout this time.

To ensure no IMP remains in the line the investigators will flush it with 50ml of sodium chloride 0.9% w/v upon completion. Volunteers will be observed for 6 hours post infusion.

Participants will be monitored during the infusion and vital signs will be recorded. Vital signs will be evaluated using a study specific Early Warning Score system.

In case of a medical emergency (e.g. anaphylaxis) infusion will be stopped immediately and action will be taken in accordance with national guidance from the UK Resuscitation Council.

There will be a delay of at least 4 hours between volunteer doses and escalation to the higher dose will not occur until 2 week safety data of the lower dose cohort has been reviewed by the trial management group. The maximum number of participants receiving IMP infusion per day will be two.

Subsequent assessments:

Serum will be collected for immunogenicity at screening, time 0 (baseline), 1, 2, 6, 24 and 48 hours, 2, 4, 8 and 12 weeks and weekly for 12 weeks.

Time 0 is defined as start of infusion. Adverse events will be assessed during the enrolment visit following the infusion and at every visit thereafter. Routine laboratory safety parameters and urine will be collected at screening, immediately post infusion and during the follow up period. ECG and vital signs will be monitored throughout the study, Volunteers will be asked to complete a diary card up to 2 weeks post-injection. Clear instruction will be provided during the immunisation visit.

Additional visits:

Additional visits and assessments may be required to evaluate an adverse event, and/or identify a diagnosis.

Referral to an independent specialist with the appropriate expertise will be arranged if there is uncertainty about the causal relationship to the IMP.

Data will be recorded directly onto the participant's medical notes or where these do not exist in the participant's trial notes and the CRFs in the most logical order.

Safety information will be collected and reported as per GCP, casualty assessment of all adverse events in relation to the IMP will also take place.

All data will be handled in accordance with the Data Protection Act 1998.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged between 18 and 45 years on the day of screening
2. Available for follow-up for the duration of the study
3. Willing and able to give written informed consent
4. At low risk of HIV and willing to remain so for the duration of the study defined as:

   1. no history of injecting drug use in the previous ten years
   2. no gonorrhoea or syphilis in the last six months
   3. no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months
   4. no unprotected anal intercourse in the last six months, outside a relationship with a regular partner known/presumed to be HIV negative
   5. no unprotected vaginal intercourse in the last six months outside a relationship with a regular known/presumed HIV negative partner
5. Willing to undergo a HIV test
6. If sexually active, using an effective method of contraception with partner (combined oral contraceptive pill; injectable or implanted contraceptive; any IUCD/IUS; consistent record with condoms if using these; physiological or anatomical sterility in self or partner) from 14 days prior to the first infusion until 4 months after, and willing to undergo urine pregnancy tests as per schedule
7. Agree to abstain from donating blood for three months after the end of their participation in the trial, or longer if necessary
8. Registered with a GP
9. Satisfactory response received from GP before randomisation

Exclusion Criteria:

1. Pregnant or lactating
2. Clinically relevant abnormality on history or examination including

   1. history of grand-mal epilepsy
   2. skin disorder might prevent insertion of IV line
   3. liver disease with inadequate hepatic function (grade 1 or greater as described in appendix 3)
   4. haematological, metabolic, gastrointestinal or cardio-pulmonary disorders
   5. uncontrolled infection; immunodeficiency or use of immunosuppressives in preceding 3 months (including systemic steroids for longer than 14 days)
   6. history of renal disease
   7. history of autoimmune disease
3. Known hypersensitivity to any component of the infusion used in this trial, or have severe or multiple allergies to drugs or pharmaceutical agents
4. History of severe local or general reaction to vaccination which according to the investigators judgement might prevent participation
5. Receipt of blood products or immunoglobulin within 4 months of screening
6. Participation in another trial of a medicinal product, completed less than 30 days prior to enrolment
7. HIV 1/2 positive or indeterminate on screening
8. Positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
9. A clinically significant amount of protein or blood in the urine
10. Grade 1 or above routine laboratory parameters (see appendix 3 for definitions). Hyperbilirubinemia to be considered an exclusion criterion only when confirmed to be conjugated bilirubinaemia
11. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
12. Unlikely to comply with protocol or the PI has any concerns about suitability of participation in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events and serious adverse events assessed by CTCAE v4.0. | three months
Number of participants with local and systemic reactogenicity signs and symptoms post-infusion | three months

SECONDARY OUTCOMES:
Serum concentration of P2G12 in participants in the active study cohorts | three months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cosgrove, Principal Investigator — St George's, University of London
Locations (1):
- St George's NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mascola JR, Montefiori DC. The role of antibodies in HIV vaccines. Annu Rev Immunol. 2010;28:413-44. doi: 10.1146/annurev-immunol-030409-101256. PMID 20192810
- [Result] Klein F, Mouquet H, Dosenovic P, Scheid JF, Scharf L, Nussenzweig MC. Antibodies in HIV-1 vaccine development and therapy. Science. 2013 Sep 13;341(6151):1199-204. doi: 10.1126/science.1241144. PMID 24031012
- [Result] Mascola JR, Haynes BF. HIV-1 neutralizing antibodies: understanding nature's pathways. Immunol Rev. 2013 Jul;254(1):225-44. doi: 10.1111/imr.12075. PMID 23772623
- [Result] Mascola JR, Stiegler G, VanCott TC, Katinger H, Carpenter CB, Hanson CE, Beary H, Hayes D, Frankel SS, Birx DL, Lewis MG. Protection of macaques against vaginal transmission of a pathogenic HIV-1/SIV chimeric virus by passive infusion of neutralizing antibodies. Nat Med. 2000 Feb;6(2):207-10. doi: 10.1038/72318. PMID 10655111
- [Result] Armbruster C, Stiegler GM, Vcelar BA, Jager W, Michael NL, Vetter N, Katinger HW. A phase I trial with two human monoclonal antibodies (hMAb 2F5, 2G12) against HIV-1. AIDS. 2002 Jan 25;16(2):227-33. doi: 10.1097/00002030-200201250-00012. PMID 11807307
- [Result] Armbruster C, Stiegler GM, Vcelar BA, Jager W, Koller U, Jilch R, Ammann CG, Pruenster M, Stoiber H, Katinger HW. Passive immunization with the anti-HIV-1 human monoclonal antibody (hMAb) 4E10 and the hMAb combination 4E10/2F5/2G12. J Antimicrob Chemother. 2004 Nov;54(5):915-20. doi: 10.1093/jac/dkh428. Epub 2004 Sep 29. PMID 15456731
- [Result] Ledgerwood JE, Coates EE, Yamshchikov G, Saunders JG, Holman L, Enama ME, DeZure A, Lynch RM, Gordon I, Plummer S, Hendel CS, Pegu A, Conan-Cibotti M, Sitar S, Bailer RT, Narpala S, McDermott A, Louder M, O'Dell S, Mohan S, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Mascola JR, Graham BS; VRC 602 Study Team. Safety, pharmacokinetics and neutralization of the broadly neutralizing HIV-1 human monoclonal antibody VRC01 in healthy adults. Clin Exp Immunol. 2015 Dec;182(3):289-301. doi: 10.1111/cei.12692. Epub 2015 Sep 24. PMID 26332605
- [Result] Mehandru S, Vcelar B, Wrin T, Stiegler G, Joos B, Mohri H, Boden D, Galovich J, Tenner-Racz K, Racz P, Carrington M, Petropoulos C, Katinger H, Markowitz M. Adjunctive passive immunotherapy in human immunodeficiency virus type 1-infected individuals treated with antiviral therapy during acute and early infection. J Virol. 2007 Oct;81(20):11016-31. doi: 10.1128/JVI.01340-07. Epub 2007 Aug 8. PMID 17686878
- [Result] Trkola A, Kuster H, Rusert P, Joos B, Fischer M, Leemann C, Manrique A, Huber M, Rehr M, Oxenius A, Weber R, Stiegler G, Vcelar B, Katinger H, Aceto L, Gunthard HF. Delay of HIV-1 rebound after cessation of antiretroviral therapy through passive transfer of human neutralizing antibodies. Nat Med. 2005 Jun;11(6):615-22. doi: 10.1038/nm1244. Epub 2005 May 8. PMID 15880120
- [Result] Ma JK, Drossard J, Lewis D, Altmann F, Boyle J, Christou P, Cole T, Dale P, van Dolleweerd CJ, Isitt V, Katinger D, Lobedan M, Mertens H, Paul MJ, Rademacher T, Sack M, Hundleby PA, Stiegler G, Stoger E, Twyman RM, Vcelar B, Fischer R. Regulatory approval and a first-in-human phase I clinical trial of a monoclonal antibody produced in transgenic tobacco plants. Plant Biotechnol J. 2015 Oct;13(8):1106-20. doi: 10.1111/pbi.12416. Epub 2015 Jul 3. PMID 26147010
- [Result] UNAIDS Fact sheet 2015
- [Result] WHO Global Health Observatory